CLINICAL TRIAL: NCT03062514
Title: Vagus Nerve Stimulation for Pediatric Intractable Epilepsy (VNS-PIE)
Brief Title: Trial to Evaluate the Safety and Effectiveness of Vagus Nerve Stimulation for Children With Refractory Epilepsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-026
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-02

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Subjects'Vagus Nerve stimulator is on always
  Interventions: Device: PINS Vagus Nerve Stimualtor
- Control (Sham Comparator): Subjects'Vagus Nerve stimulator is off from enrollment to 3 month
  Interventions: Device: PINS Vagus Nerve Stimualtor

INTERVENTIONS:
Device: PINS Vagus Nerve Stimualtor — PINS Vagus Nerve Stimualtor

SUMMARY:
Children with refractory epilepsy who are candidates for a treatment with vagus nerve stimulation will be prospectively randomized into 2 arms. Vagus nerve stimulation parameters are programmed and adjusted during outpatient clinic visits, within the normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-6
2. At least 6 seizure per month
3. Refractory Epilepsy
4. In good health except epilepsy
5. Patients or his(her) familyscould understand this method and sign the informed consent
6. Patients with good compliance and could complete postoperative follow-up

Exclusion Criteria:

1. Results of MRI remind epilepsy caused by intracranial space-occupying lesions
2. The vagus nerve lesion and damage
3. Tumor, cardiopulmonary anomaly, progressive neurological diseases, asthma，mental disease，pepticulcer，diabetes，bad health etc, and other surgical contraindication
4. Cann't write the epilepsy diary
5. Participating other clinical trial
6. Cann't complate the operation
7. Complete the postoperative follow-up
8. Cann't complete the promgramming

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in seizure frequency | 12 weeks of stimulation

SECONDARY OUTCOMES:
Changes in seizure frequency | 6、12、24 weeks of stimulation
Engel scale description | 6、12、24 weeks of stimulation
Changes in the Number of Anti-epileptic Drugs | 6、12、24 weeks of stimulation
GESELL mental development scales | 12、24 weeks of stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Yuwu Jiang, MD, Principal Investigator — Peking University First Hospital; Liping Zou, Study Director — Chinese PLA General Hospital; Jianxiang Liao, Study Director — Shenzhen Children's Hospital; Qian Chen, Study Director — Children's Hospital of The Capital Institute of Pediatrics; Baomin Li, Study Director — Qilu Hospital of Shandong University; Yuxing Gao, Study Director — Shandong Provincial Hospital; Jianmin Liang, Study Director — The First Hospital of Jilin University; Shaoping Huang, Study Director — Second Affiliated Hospital of Xi'an Jiaotong University; Fei Yin, Study Director — Xiangya Hospital of Central South University; Feng Gao, Study Director — The Children's Hospital of Zhejiang University School of Medicine; Yanhui Chen, Study Director — Fujian Medical University Union Hospital; XiaoMei SHU, Study Director — Zunyi Medical College; Hua Yu, Study Director — Shengjing Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Panebianco M, Rigby A, Marson AG. Vagus nerve stimulation for focal seizures. Cochrane Database Syst Rev. 2022 Jul 14;7(7):CD002896. doi: 10.1002/14651858.CD002896.pub3. PMID 35833911
- [Derived] Ji T, Yang Z, Liu Q, Liao J, Yin F, Chen Y, Zou L, Li B, Gao Y, Shu X, Huang S, Gao F, Liang J, Lin SF, Peng J, Song S, Wang J, Che C, Sun W, Tian M, Yang L, Hua Y, Hao Y, Cai L, Li L, Jiang Y. Vagus nerve stimulation for pediatric patients with intractable epilepsy between 3 and 6 years of age: study protocol for a double-blind, randomized control trial. Trials. 2019 Jan 14;20(1):44. doi: 10.1186/s13063-018-3087-4. PMID 30642370